CLINICAL TRIAL: NCT01819090
Title: Optimizing Communication During Nasal Mechanical Ventilation
Brief Title: Optimizing Communication During Ventilation
Acronym: PHONOVNI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Principal Investigator, Helene Prigent, MDPHD, Centre d'Investigation Clinique et Technologique 805
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012- A01394-39
Record Dates: First submitted 2013-03-07; First posted 2013-03-27 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2015-10

CONDITIONS: Neuromuscular Disorder; Respiratory Failure
Keywords: Neuromuscular disorder; Mechanical ventilation; Speech; Respiratory failure
MeSH Terms: conditions — Neuromuscular Diseases; Respiratory Insufficiency; Speech

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No ventilation switch control (Active Comparator): Neuromuscular patients non invasively ventilated in a stable state at the time of the study testing an usual (with no ventilation switch control) Elysee 150 ventilator while speaking
  Interventions: Device: Elysee 150 ventilator
- Ventilation switch control (Active Comparator): Neuromuscular patients non invasively ventilated in a stable state at the time of the study testing an Elysee 150 ventilator with a ventilation switch control allowing them to control ventilation while speaking
  Interventions: Device: Elysee 150 ventilator with a ventilation switch control

INTERVENTIONS:
Device: Elysee 150 ventilator
  Other Names: Elysee 150 - Resmed
  Arms: No ventilation switch control
Device: Elysee 150 ventilator with a ventilation switch control
  Other Names: Elysee 150 ventilator - Resmed - with a ventilation switch control
  Arms: Ventilation switch control

SUMMARY:
Mechanical ventilation is one of the only treatment that has improved survival of patients with neuromuscular respiratory failure. As disease progresses, some patients may require longer ventilation period. Non invasive mechanical ventilation is the preferred method of ventilation but it may interfere with speech and communication of patients who require ventilation throughout the day. The investigators are evaluating the effect on speech and communication of a ventilation device which allows patients to momentarily and voluntarily withhold ventilation if they want to speak. This should allow the patients to have a more fluid speech.

ELIGIBILITY:
Inclusion Criteria:

* Patient with restrictive respiratory failure secondary to a neuromuscular disorder, without any bulbar involvement.
* Age greater than or equal to 18.
* Hospitalization in Home Ventilation Unit of the intensive care department of R. Poincaré Hospital.
* Non invasive mechanical ventilation for a duration equal or above 14h per day.
* Patient in a steady state at the time of the study
* written informed consent

Exclusion Criteria:

* patient's refusal to participate to the study
* Inability to read the selected text
* Inability to use the ventilator switch
* Inability to cooperate
* Hemodynamic instability
* Acute respiratory failure
* No affiliation to social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Impact of patient's ventilation control on speech efficiency | 1 hour 30 min
  Speech efficiency will be evaluated while using a ventilator which allows the patient to constantly control when he wants to be ventilated Speech evaluation is based on speech rhythm and text reading duration

SECONDARY OUTCOMES:
Patient ventilator synchronisation during speech | 1hour 30 min
  Evaluated with the variation of respiratory frequency during speech, the number of auto-triggered ventilation cycles during speech.
User friendliness of the ventilator during speech | 1hour 30 min
  evaluation of user friendliness by the patient using a visual analogical score
Respiratory comfort during speech | 1hour 30 min
  evaluation of user friendliness by the patient using a visual analogical score and the Borg score
Speech comfort during ventilation | 1hour 30 min
  evaluation of speech comfort during ventilation by the patient using a visual analogical score

CONTACTS AND LOCATIONS:
Overall Officials: Helene PRIGENT, MDPHD, Principal Investigator — Hôpital RAYMOND POINCARE
Locations (1):
- Hopital Raymond Poincare, Garches, Garches, France